CLINICAL TRIAL: NCT06183801
Title: GLAC Metabolic Regulatory Probiotics, the Evaluation to Improve the Human Metabolic Syndrome, Intestinal Microflora and Short Chain Fatty Acid.
Brief Title: Effects of Probiotics on Metabolic Syndrome ,Intestinal Microflora and SCFA.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glac Biotech Co., Ltd (Industry)
Responsible Party: Principal Investigator, Hsieh-Hsun Ho, R & D director, Glac Biotech Co., Ltd
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: FYH-IRB-110-01-02
Record Dates: First submitted 2023-12-04; First posted 2023-12-28 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Metabolic Syndrome
Keywords: Probiotics; Gut microbiota; Metabolic imbalances; SCFAs
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Probiotic 1 (Experimental): Subjects take probiotics capsule three times a day before meal.
  Interventions: Dietary Supplement: Probiotics 1
- Probiotic 2 (Experimental): Subjects take probiotics capsule three times a day before meal.
  Interventions: Dietary Supplement: Probiotics 2
- Probiotic 3 (Experimental): Subjects take probiotics capsule three times a day before meal.
  Interventions: Dietary Supplement: Probiotics 3
- Probiotic 4 (Experimental): Subjects take probiotics capsule three times a day before meal.
  Interventions: Dietary Supplement: Probiotics 4
- Probiotic 5 (Experimental): Subjects take probiotics capsule three times a day before meal.
  Interventions: Dietary Supplement: Probiotics 5
- Placebo 1 (Placebo Comparator): Subjects take probiotics capsule three times a day before meal.
  Interventions: Dietary Supplement: Placebo 1
- Probiotic 6 (Experimental): After 1 month wash out,subjects take probiotics capsule three times a day before meal.
  Interventions: Dietary Supplement: Probiotics 6
- Probiotic 7 (Experimental): After 1 month wash out,subjects take probiotics capsule three times a day before meal.
  Interventions: Dietary Supplement: Probiotics 7
- Placebo 2 (Placebo Comparator): After 1 month wash out,subjects take probiotics capsule three times a day before meal.
  Interventions: Dietary Supplement: Placebo 2

INTERVENTIONS:
Dietary Supplement: Probiotics 1 — Subjects take probiotics capsule(Lactobacillus fermentum,TSF331) three times a day before meal.
  Arms: Probiotic 1
Dietary Supplement: Probiotics 2 — Subjects take probiotics capsule(Lactobacillus reuteri,TSR332) three times a day before meal.
  Arms: Probiotic 2
Dietary Supplement: Probiotics 3 — Subjects take probiotics capsule(Lactobacillus plantarum,TSP05) three times a day before meal.
  Arms: Probiotic 3
Dietary Supplement: Probiotics 4 — Subjects take probiotics capsule(Lactobacillus fermentum,TSF331+Lactobacillus reuteri,TSR332+Lactobacillus plantarum,TSP05) three times a day before meal.
  Arms: Probiotic 4
Dietary Supplement: Probiotics 5 — Subjects take probiotics capsule(Lactobacillus fermentum,TSF331+Lactobacillus reuteri,TSR332+Lactobacillus plantarum,TSP05+Postbiotics PE0401) three times a day before meal.
  Arms: Probiotic 5
Dietary Supplement: Placebo 1 — Subjects take capsule three times a day before meal.
  Arms: Placebo 1
Dietary Supplement: Probiotics 6 — After 1 month wash out, subjects take probiotics capsule(Bifidobacterium animalis subsp. lactis,CP-9) three times a day before meal.
  Arms: Probiotic 6
Dietary Supplement: Probiotics 7 — After 1 month wash out, subjects take probiotics capsule(Lactobacillus rhamnosus, bv-77+Bifidobacterium animalis subsp. lactis,CP-9) three times a day before meal.
  Arms: Probiotic 7
Dietary Supplement: Placebo 2 — After 1 month wash out, subjects take capsule three times a day before meal.
  Arms: Placebo 2

SUMMARY:
The improvement effects of GLAC biotech probiotics contains 5 specialized strains on the biochemical analysis and gut microbiota will be verified in the clinical trial through cooperation with the ADPRC. Through this project, the difference and improvement before and after the GLAC biotech probiotics taking will be clinically validated fromseveral aspects, including blood biochemical values, NGS gut microbiota analysis, GAIS and SCFAs levels. Therefore, by this industry- academic cooperation project, the investigators can explore the improvement of human gut microbiota by GLAC biotech probiotics, to understand the essence of clinical benefit, and the investigators expect the accomplishments of this project can help the consumers understand the added value and excellence of the GLAC products, and thus enhance consumer confidence and expand product markets.

DETAILED DESCRIPTION:
In recent years, the issue of gut microbiota and probiotics has been becoming very popular, and more and more gastrointestinal health foods have been developed and commercialized. The impact of gut microbiota on human health has received increasing attention and expectations from the world. Probiotics are one of the most recognized and positive health materials for consumers. Lactobacillus/probiotics, the main raw materials of health foods most frequently purchased by domestic consumers in recent years, have always ranked the first. They have certain improvement effects in terms of gastrointestinal improvement, immune regulation, and blood lipid regulation. There are currently about 30 probiotic manufacturers in Taiwan. Since the regulations do not have any clinical functional requirements for probiotic products, most probiotic products only describe the characteristics, functions and animal experiments of probiotics. There is no actual clinical experimental data to verify the effect of probiotic products on human intestinal flora. The probiotics researched and developed by GLAC Biotechnology company have undergone rigorous in vitro and animal tests, and actively cooperate with domestic and foreign hospitals to conduct human clinical trials to verify the function of the strains.

With the progress of human culture and lifestyle, many diseases of modern civilization have emerged one after another. Most of these diseases are caused by changes of lifestyle or diet, leading to the human body's metabolic imbalances, such as high blood sugar, high cholesterol, hypertension, hyperuricemia, liver dysfunction, and obesity. Gut dysbiosis and diseases associated with aging usually have such phenomenon like increased pathogenic bacteria, decreased probiotics decrease and declined gut microbiota diversity. The gut dysbiosis contributes to the aging gut and aging-related diseases in at least three aspects including production of Lipopolysaccharides (LPS), reduced levels of short chain fatty acids (SCFAs), and inflamm-aging. The next generation sequencing (NGS) technology can provide high throughput, high sensitivity and reliable detection, and then the investigators can understand improving effects of the human gut microbiota. The Aging and Disease Prevention Research Center (ADPRC) of the Fooyin university has a complete and skilled next generation sequencing (NGS) platform and a gut microbiota database included 5000 clinical cases, and thus provide the best clinical verification platform for probiotic products. Based on the common probiotic/pathogenic markers, reported in most of studies, and 4 specific domestic markers found in our study, the investigators have defined the domestic gut aging index score (GAIS) to predict the aging of the gut. The GASI provides an excellent discrimination. In addition, gut microbiota normally affects inflammatory cytokines by generating SCFAs to modulate the immune system against pathogens. The improvement effects of GLAC biotech probiotics contains 5 specialized strains on the biochemical analysis and gut microbiota will be verified in the clinical trial through cooperation with the ADPRC. Through this project, the difference and improvement before and after the GLAC biotech probiotics taking will be clinically validated from several aspects, including blood biochemical values, NGS gut microbiota analysis, GAIS and SCFAs levels. Therefore, by this industry- academic cooperation project, the investigators can explore the improvement of human gut microbiota by GLAC biotech probiotics, to understand the essence of clinical benefit, and the investigators expect the accomplishments of this project can help the consumers understand the added value and excellence of the GLAC products, and thus enhance consumer confidence and expand product markets.

ELIGIBILITY:
Inclusion Criteria:

1. The subject are willing to provide physical examination reports within the past 1 year.
2. The subject are willing to sign informed consent form.

Exclusion Criteria:

1. Pregnant women or preparing for pregnancy.
2. The subject were taking antibiotics.
3. One of parents are not Han Chinese or aboriginal.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
blood biochemical indicators | Day0、Day30、Day60、Day90、Day120、Day180
  Detecting the changes of concentration in blood biochemical indexes .
  1. glucose AC (mg/dL)
  2. Glutamic Oxaloacetic Transaminase,GOT (U/L)
  3. Glutamic Pyruvic Transaminase,GPT (U/L)
  4. Blood urea nitrogen,BUN (mg/dL)
  5. Creatinine (mg/dL)
  6. Triglyceride,TG (mg/dL)
  7. total cholesterol (mg/dL)
  8. High-density lipoprotein,HDL (mg/dL)
  9. Low-density lipoprotein,LDL (mg/dL)
Changes in gut microbiota ratios | Day0、Day30、Day60、Day90、Day120、Day180
  Using Next-Generation Sequencing (NGS) to analyze the changes of fecal flora.
Changes in gut aging index score(GAIS) | Day0、Day30、Day60、Day90、Day120、Day180
  Calculating probiotic/pathogenic ratios

SECONDARY OUTCOMES:
Short chain fatty acid analysis | Day0、Day30、Day60、Day90、Day120、Day180
  Changerate of short chain fatty acid in stool
Changes in sleep quality | Day0、Day30、Day60、Day90、Day120、Day180
  PITTSBURGH SLEEP QUALITY INDEX (PSQI):The minimum value is "0" and maximum value is "72", higher scores mean a worse outcome.
  The change in score will be evaluated.
Evaluating the score difference of Gastrointestinal(GI) symptoms questionnaire | Day0、Day30、Day60、Day90、Day120、Day180
  Gastrointestinal(GI) symptoms questionnaire:The minimum value is "0" and maximum value is "30", higher scores mean a worse outcome.The change in score will be evaluated.
Evaluating the score difference of Physical symptoms questionnaire | Day0、Day30、Day60、Day90、Day120、Day180
  Physical symptoms questionnaire:The minimum value is "0" and maximum value is "75", higher scores mean a worse outcome.The change in score will be evaluated.
Changes in stool form | Day0、Day30、Day60、Day90、Day120、Day180
  Record the stool form and color.Types 1 and 2 indicate constipation, with 3 and 4 being the ideal stools as they are easy to defecate while not containing excess liquid, 5 indicating lack of dietary fiber, and 6 and 7 indicate diarrhoea.(Type 1: Separate hard lumps, like nuts (difficult to pass)、Type 2: Sausage-shaped, but lumpy、Type 3: Like a sausage but with cracks on its surface、Type 4: Like a sausage or snake, smooth and soft (average stool)、Type 5: Soft blobs with clear cut edges、Type 6: Fluffy pieces with ragged edges, a mushy stool (diarrhea)、Type 7: Watery, no solid pieces, entirely liquid (diarrhea))

CONTACTS AND LOCATIONS:
Overall Officials: Hsieh-Hsun Ho, Ph. D., Principal Investigator — Study Principal Investigator
Locations (1):
- Glac Biotech Co., Ltd., Tainan, Taiwan

REFERENCES:
- [Derived] Lin JH, Lin CH, Kuo YW, Liao CA, Chen JF, Tsai SY, Li CM, Hsu YC, Huang YY, Hsia KC, Yeh YT, Ho HH. Probiotic Lactobacillus fermentum TSF331, Lactobacillus reuteri TSR332, and Lactobacillus plantarum TSP05 improved liver function and uric acid management-A pilot study. PLoS One. 2024 Jul 24;19(7):e0307181. doi: 10.1371/journal.pone.0307181. eCollection 2024. PMID 39046973